CLINICAL TRIAL: NCT05477017
Title: Prospective Observational Cohort Study to Evaluate the Benefits, Documented in the Experimental Settings, of Treatment With SGLT2-i in Normal Clinical Practice, in Subjects With Type 2 Diabetes and Older Than 70 Years.
Brief Title: Evaluation of SGLT2-i Effectivness and Safety in Elderly Type 2 Diabetes Patients
Acronym: SOLDMiDiab02
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Principal Investigator, University of Milan
Other Study IDs: 03/2022
Record Dates: First submitted 2022-05-23; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Type2Diabetes
Keywords: SGLT2-inhibitors; Elderly; Safety
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; dapagliflozin; Canagliflozin; ertugliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: SGLT2 inhibitor — Selective inhibitors of the sodium and glucose co-transporter 2 (SGLT2) originated as antidiabetic drugs thanks to their hypoglycemic and glycosuric effect.
  Other Names: Jardiance; Synjardy; Forxiga; Xigduo; Invokana; Vokanamet; Steglatro; Segluromet

SUMMARY:
The aim of the study is to evaluate the benefits, documented in experimental settings, of treatment with SGLT2-i in subjects with type 2 diabetes and older than 70 years in normal clinical practice.

The type of study does not involve immediate risks or direct benefits for the subjects taking part in it. The potential benefits for clinicians and healthcare systems are: greater knowledge of diabetic disease and the study of new treatment options. However, the analysis of the data will allow us to better identify which patients benefit most from treatment with glycosurics.

DETAILED DESCRIPTION:
Sodium-glucose co-transporter-2 inhibitors (SGLT2i) may have important benefits for the elderly with type 2 diabetes (T2D), however some safety concerns still limit their use in patients over 70 years of age. The SOLD study (SGLT2-i in Older Diabetic patients) aim to evaluate which basal characteristics of the patients are more frequently related to the suspension of treatment with SGLT2-i in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent issued before any other activity related to the study (i.e. any activity related to data collection according to the study protocol);
* Diagnosis of type II diabetes mellitus, according to ADA indications for at least 3 months
* Males or females > 70 years old
* Stable therapy for at least 3 months with oral hypoglycemic agents / insulin
* Prescription of SGLT2 inhibitors, in accordance with normal clinical practice and local drug prescription / reimbursement guidelines.

Exclusion Criteria:

* Mental incapacity, unavailability or language barriers that preclude adequate understanding or cooperation;
* Diagnosis of type 1 diabetes mellitus, MODY (maturity-onset diabetes of the young), LADA (latent autoimmune diabetes in adults), gestational diabetes mellitus, secondary diabetes mellitus or any other hyperglycemic state other than T2D;
* Previous participation in the study. Participation is defined by having given informed consent to the study;
* Participation in another clinical study on T2D that includes any clinical intervention or administration of an investigational drug within 3 months prior to enrollment in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly with type 2 diabetes receiving SGLT2-i therapy
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Variation in HbA1c values (% -point) | From Baseline to 12 months
  Variation in HbA1c values (% -point) from baseline to 12 months from enrollment

SECONDARY OUTCOMES:
Evaluation of the maintenance of glycemic compensation | From Baseline to 12 months
  Evaluation of the maintenance of glycemic compensation after the initiation of glycosuric therapy in clinical practice
Evaluation of fasting glycemic control | From Baseline to 12 months
  Evaluation of fasting glycemic control (mg/dl)
Evaluation of the weight | From Baseline to 12 months
  Evaluation of the weight (Kg)
Evaluation of the BMI | From Baseline to 12 months
  Evaluation of the BMI (Kg/m2)
Evaluation of the waist circumference | From Baseline to 12 months
  Evaluation of the waist circumference (cm)
Evaluation of the systolic and diastolic pressure | From Baseline to 12 months
  Evaluation of the systolic and diastolic pressure (mmHg)
Evaluation of the heart rate | From Baseline to 12 months
  Evaluation of the heart rate (bpm)
Evaluation of the serum creatinine | From Baseline to 12 months
  Evaluation of the serum creatinine (mg/dl)
Evaluation of the e-GFR | From Baseline to 12 months
  Evaluation of the e-GFR (mL/min/1.73m2)
Evaluation of the main side effects and the withdrawal rate | From Baseline to 12 months
  Evaluation of the main side effects and the withdrawal ratein the first year of treatment. It will be evalueted through scheduled clinical visit

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, Principal Investigator — ASST FBF-Sacco
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Diabetes Association. 12. Older Adults: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S139-S147. doi: 10.2337/dc19-S012. PMID 30559238
- [Result] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Result] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Result] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Result] Pham SV, Chilton RJ. EMPA-REG OUTCOME: The Cardiologist's Point of View. Am J Cardiol. 2017 Jul 1;120(1S):S53-S58. doi: 10.1016/j.amjcard.2017.05.011. Epub 2017 May 30. PMID 28606345
- [Result] Cahn A, Mosenzon O, Wiviott SD, Rozenberg A, Yanuv I, Goodrich EL, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS, Raz I. Efficacy and Safety of Dapagliflozin in the Elderly: Analysis From the DECLARE-TIMI 58 Study. Diabetes Care. 2020 Feb;43(2):468-475. doi: 10.2337/dc19-1476. Epub 2019 Dec 16. PMID 31843945